CLINICAL TRIAL: NCT05314218
Title: EPICADIA - Electrophysiologic Performance Investigation for CArdiac DIAgnosis
Brief Title: The Objective of This Multicentre Study is to Collect Operative Data on the Related Clinical Functional Outcomes and Complications and of Market Approved Alcis Electrophysiology Catheters to Demonstrate Safety and Performance of These Devices in a Real-world Setting
Status: Completed | Type: Observational
Sponsor: Alcis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2045-CIP_v1_01Feb2022
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Electrophysiology catheters and cables — The Xtrem electrophysiology catheter was developed for diagnosis of cardiac arrhythmias. Their function is to collect by contact, electrical signals generated by the heart muscle.
  Xtrem are inserted via femoral vena cava or via artery and can be used in two occasions:
  * Exploration procedures for diagnosis alone
  * Diagnosis before ablation procedure An extension cable is used to connect the catheter to a stimulation/ recording device.

SUMMARY:
The objective of this multicentre study is to collect operative data on the related clinical functional outcomes and complications and of market approved Alcis electrophysiology catheters to demonstrate safety and performance of these devices in a real-world setting.

DETAILED DESCRIPTION:
Outcome data collected from this study will provide the basis for Post-Market Surveillance (PMS) reporting, Clinical Study Report (CSR), Clinical Evaluation Report (CER) on Alcis devices and support peer-reviewed publications on products performance and safety.

ELIGIBILITY:
Inclusion Criteria:

To be included, patients must be:

* 18 to 90 years old
* Patient who have to undergo diagnostic procedure or ablation procedure (Cardiac arrythmias)
* Informed and willing to sign an informed consent for approved by EC
* Affiliation to the social security or foreign regime recognized in France

Exclusion Criteria:

A patient will not be eligible to participate in the study if any of the following conditions are present:

* Not able to comply with the study procedures based on the judgment of the assessor (e.g. cannot comprehend study questions, inability to keep scheduled assessment times).
* Any medical condition that could impact the study at investigator's discretion (e.g. allergy…).
* Pregnant women
* Adult subject to legal protection measure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have to undergo diagnostic procedure or ablation procedure (Cardiac arrythmias).
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Signal quality | Through study completion, an average of 4 hours
  Good signal amplitude and signal stability throughout the procedure without artefact

SECONDARY OUTCOMES:
Micro-stimulation | Through study completion, an average of 4 hours
  Micro-stimulation worked well.
Manoeuvrability | Through study completion, an average of 4 hours
  Ease of positioning and manoeuvrability the catheter (access to the desired area)
Bending | Through study completion, an average of 4 hours
  Link between the wheel and the bending for dynamic Xtrem and bending stability
Imaging | Through study completion, an average of 4 hours
  Visibility via X ray or 3D navigation.
Diagnosis | Through study completion, an average of 4 hours
  Diagnosis efficiency

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Rhône Durance, Avignon
  - Hôpital Henri-Mondor AP-HP, Créteil, Île-de-France Region